CLINICAL TRIAL: NCT01085149
Title: The Effect Of Simvastatin On Bone Remodeling In Socket Of Mandibular Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: dr. casap nardi, hadassah medical organization, jerusalem, israel
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: h123-HMO-CTIL
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Hypercholesterolemia
Keywords: simvastatin; alveolar bone; tooth extraction; remodeling; alveolar bone remodeling
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): simvastatin will be inserted to sockets
  Interventions: Drug: Simvastatin
- control (No Intervention): sockets will be left to healing without material in socket
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 10 mg simvastatin, slow release in socket of extracted tooth (single application only)

SUMMARY:
Simvastatin has been reported to promote osteoblastic activity and inhibit osteoclastic activity by enhancing the expression of BMP2. There have been many studies demonstrating the bone-promoting effect of local application various animal models including after application into socket of teeth in a rat. the purpose of the study is to investigate the effect of slow release topical simvastatin in socket of mandibular teeth on bone remodeling in the socket

DETAILED DESCRIPTION:
after extraction of mandibular single root teeth 10 mg of slow release simvastatin would be inserted to the socket. observation will be at 1 week, 4 weeks and 3 months.after 3 months the patients will have dental CT as done routinely in our clinic before placing dental implants and the bone density and height will be measured on this data. during the procedure of inserting a dental implant a trephine will be taken for histology.

ELIGIBILITY:
Inclusion Criteria:

* need extraction of single root tooth
* intend to have prosthetic implant in place of extraction

Exclusion Criteria:

* treated with simvastatin P.O for hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
bone height and density in former socket | 3 months
  measured on CT

SECONDARY OUTCOMES:
bone mineralization | 3 months
  histology from bone in former socket

CONTACTS AND LOCATIONS:
Overall Officials: casap nardi, MD, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Oral and Maxillofacial Clinic, Hadassah, Jerusalem, Israel

REFERENCES:
- [Background] Wu Z, Liu C, Zang G, Sun H. The effect of simvastatin on remodelling of the alveolar bone following tooth extraction. Int J Oral Maxillofac Surg. 2008 Feb;37(2):170-6. doi: 10.1016/j.ijom.2007.06.018. Epub 2007 Sep 4. PMID 17804200